CLINICAL TRIAL: NCT03281668
Title: Feasibility of High Intensity Interval Training in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-2996; 1R21HD088852-01A1 (NIH)
Record Dates: First submitted 2017-08-31; First posted 2017-09-13 (Actual); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Single Group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Intervention consists of High Intensity Interval Training (HIIT) session which is af 3-5 minute warm up, followed by 10 repetitions of 1 minute bouts at individualized training intensity with 1 minute rest periods.
  Interventions: Behavioral: High intensity interval training (HIIT)

INTERVENTIONS:
Behavioral: High intensity interval training (HIIT) — Each training session for High Intensity Interval Training will consist of a 3-5 minute warm-up, followed by 10 repetitions of 1-minute bouts at individualized training intensity with 1-minute rest periods.

SUMMARY:
The focus of this pilot study is to evaluate the feasibility of utilizing an evidenced-based high intensity interval training program (HIIT) to improve physical function in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
All participants will be assigned to the single-arm of the study in which all participants will receive 12 weeks of HIIT, delivered twice per week. The primary outcome will examine the feasibility and acceptability of the 12 week HIIT program in patients with knee OA symptoms ranging from mild to severe. The investigators will determine adherence to and tolerability of HIIT, acceptability, and recruitment and retention rates during the 12 week program. Additional outcomes will include physical function, knee OA symptomatic burden (pain), static standing balance, isometric knee extensor and flexor strength, cardiorespiratory fitness, and body composition.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 40 and 75 years old
* body mass index of 18.5-50 kg/m²
* exhibits symptomatic knee OA, defined as a diagnosis of knee OA, as identified from University of North Carolina electronic medical records, and current knee symptoms in at least one knee, having a minimum score of 6 out of 20 on the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC) pain subscale.

Exclusion Criteria:

* individuals diagnosed with a cardiovascular condition restricting exercise
* individuals currently meeting Department of Health and Human Services Guidelines for physical activity (≥ 150 minutes per week
* individuals currently doing HIIT
* individuals currently participating in physical therapy for knee OA
* individuals currently participating in another OA intervention study
* received a corticosteroid or hyaluronic acid intra-articular injection in the knee during the previous 3 weeks or scheduled for during the intervention
* diagnosis of gout in the knee
* diagnosis of rheumatoid arthritis
* diagnosis of fibromyalgia
* other systemic rheumatic disease
* severe dementia or other memory loss
* active diagnosis of psychosis or uncontrolled substance abuse disorder
* hospitalization for a stroke, heart attack, or heart failure, or had surgery for blocked arteries in the past 3 months
* total joint replacement knee surgery, other knee surgery, meniscus tear, or anterior cruciate ligament (ACL) tear in the past 6 months
* on a waiting list for total joint replacement
* severely impaired hearing or speech
* pregnant or planning to become pregnant while enrolled in the study
* inability to speak English
* serious or terminal illness as indicated by referral to hospice or palliative care
* nursing home residence
* inability to ride a stationary bike
* any other health problems that would prohibit safe participation in the study
* EKG results EKG suggesting the individual would not be able to safely participate in this study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Golightly, PT, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 29
Completed | 21
Not Completed | 8
Not completed — Physician Decision | 1
Not completed — scheduling conflict, family circumstance | 2
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: years] | 63 [44 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.8 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Potential Participants Screened for the Study Who Are Enrolled
Description: Number of participants screened and enrolled divided by the total number of participants screened
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Groups:
- Intervention: Intervention consists of High Intensity Interval Training (HIIT) session which is a 3-5 minute warm up, followed by 10 repetitions of 1 minute bouts at individualized training intensity with 1 minute rest periods.
  High intensity interval training (HIIT): Each training session for High Intensity Interval Training will consist of a 3-5 minute warm-up, followed by 10 repetitions of 1-minute bouts at individualized training intensity with 1-minute rest periods.
Arm/Group | Intervention
Number analyzed (Participants) | 150
percentage of participants | 19.3

2. Primary Outcome: Percentage of Enrolled Participants Retained at the End of the Study
Description: Number of participants who completed the study (baseline through 12 week assessments) divided by the total number of enrolled participants with baseline assessments
Time Frame: Study completion (12 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 29
percentage of participants | 72.4

3. Secondary Outcome: Average Number of Training Sessions Completed Per Week
Description: Up to 2 training sessions were possible each week over the 12 week intervention
Time Frame: Weekly measures for 12 consecutive weeks
Measure: Mean (Standard Deviation); unit: training sessions per week
Arm/Group | Intervention
Number analyzed (Participants) | 29
training sessions per week | 1.9 (0.24)

4. Secondary Outcome: Total Number of Training Sessions Completed
Description: Total number of training sessions completed out of up to 24 sessions (2 per week over 12 weeks)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: training sessions
Arm/Group | Intervention
Number analyzed (Participants) | 29
training sessions | 19.4 (7.4)

5. Secondary Outcome: Total Number of Training Weeks Completed
Description: Total number of training weeks (up to 12 weeks possible)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Intervention
Number analyzed (Participants) | 29
weeks | 11.4 (1.47)

6. Secondary Outcome: Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Total Score From Baseline to 12 Weeks
Description: The WOMAC, a measure of lower extremity pain (5 items), stiffness (2 items), and function (17 items), will be used to measure overall symptomatic burden of knee osteoarthritis (OA). Each item is scored from 0-4 (none, slight, moderate, severe, and extreme). Items are added to calculate a total WOMAC score ranging from 0 (no problems) to 96 (extreme problems). A higher score means a worse outcome.
Time Frame: Baseline,12 weeks
Measure: Mean (95% Confidence Interval); unit: percentage change in score
Arm/Group | Intervention
Number analyzed (Participants) | 21
percentage change in score | -9.2 [-13.6 to -4.9]

7. Secondary Outcome: Change in WOMAC Pain Subscale From Baseline to 12 Weeks
Description: The WOMAC pain subscale contains 5 items about knee pain. Each item is scored from 0-4 (none, slight, moderate, severe, and extreme). Items are added to calculate a WOMAC pain score ranging from 0 (no pain) to 20 (extreme pain). A higher score means more severe pain.
Time Frame: Baseline,12 weeks
Measure: Mean (95% Confidence Interval); unit: percentage change in score
Arm/Group | Intervention
Number analyzed (Participants) | 21
percentage change in score | -1.7 [-2.8 to -0.6]

8. Secondary Outcome: Change in WOMAC Function Subscale From Baseline to 12 Weeks
Description: The WOMAC function subscale contains 17 items about knee function during daily activities. Each item is scored from 0-4 (none, slight, moderate, severe, and extreme). Items are added to calculate a WOMAC pain score ranging from 0 (no problems with function) to 68 (extreme problems with function). A higher score means worse function.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: percentage change in score
Arm/Group | Intervention
Number analyzed (Participants) | 21
percentage change in score | -6.3 [-9.6 to -3.1]

9. Secondary Outcome: Change in 20m Fast Paced Walk Test
Description: Measure of the ability to walk quickly over short distances. Participants walk at fast pace that is timed over 2 x 10m.
Time Frame: Baseline, 12 weeks
Population: Originally planned to have participants perform 40-meter walk; however, due to lab space constraints, this was altered to a 20-meter walk instead.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Intervention
Number analyzed (Participants) | 21
seconds | -1.13 [-1.61 to -0.64]

10. Secondary Outcome: Change in Number of Chair Stand Repetitions Completed
Description: Number of chair stand repetitions completed in 30 seconds
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: number of chair stands
Arm/Group | Intervention
Number analyzed (Participants) | 21
number of chair stands | 2.6 [1.8 to 3.4]

11. Secondary Outcome: Change in Stair Climb Test
Description: Time in seconds to ascend and descend a flight of stairs
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: change in seconds
Arm/Group | Intervention
Number analyzed (Participants) | 21
change in seconds | -1.42 [-2.13 to -0.71]

12. Secondary Outcome: Change in Timed Up and Go
Description: Time in seconds to rise from a chair, walk 3 m, turn, walk back to chair, and sit down
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: change in seconds
Arm/Group | Intervention
Number analyzed (Participants) | 21
change in seconds | -0.58 [-0.95 to -0.22]

13. Secondary Outcome: Change in Feet Together Stand
Description: Feet together stand for up to 10 seconds without assistive device
Time Frame: Baseline, 12 weeks
Population: All participants were able to complete Feet Together Stand at baseline and 12 weeks (no change).
Measure: Mean (95% Confidence Interval); unit: change in seconds
Arm/Group | Intervention
Number analyzed (Participants) | 21
change in seconds | 0.00 [0.00 to 0.00]

14. Secondary Outcome: Change in Semi-tandem Stand
Description: Heel of one foot placed to the side of the big toe of the other foot, for up to 10 seconds
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: change in seconds
Arm/Group | Intervention
Number analyzed (Participants) | 21
change in seconds | 0.52 [-0.18 to 1.23]

15. Secondary Outcome: Change in Tandem Stand
Description: One foot in front of the other, heel touching toe, for up to 10 seconds
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: change in seconds
Arm/Group | Intervention
Number analyzed (Participants) | 21
change in seconds | 0.39 [-0.33 to 1.11]

16. Secondary Outcome: Change in One Leg Stand
Description: One leg stand for up to 30 seconds
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: change in seconds
Arm/Group | Intervention
Number analyzed (Participants) | 21
change in seconds | 3.41 [0.26 to 6.56]

17. Secondary Outcome: Change in Cardiorespiratory Fitness
Description: Measure by peak oxygen consumption (VO2peak),to identify fitness level and evaluate cardiovascular effects. Test will establish individual training intensity.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: change in liters/minute
Arm/Group | Intervention
Number analyzed (Participants) | 21
change in liters/minute | 0.14 [0.03 to 0.24]

18. Secondary Outcome: Change in Whole Body Fat Mass
Description: fat mass in kilograms, measured with dual energy x-ray absorptiometry (DXA)
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: kilogram (kg)
Arm/Group | Intervention
Number analyzed (Participants) | 21
kilogram (kg) | -0.28 [-1.10 to 0.54]

19. Secondary Outcome: Change in Lean Body Mass
Description: lean body mass in kilograms, measured with DXA
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: kilogram (kg)
Arm/Group | Intervention
Number analyzed (Participants) | 21
kilogram (kg) | -0.12 [-0.56 to 0.31]

20. Secondary Outcome: Change in Visceral Fat
Description: visceral fat in kilograms, measured with DXA
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: kilogram (kg)
Arm/Group | Intervention
Number analyzed (Participants) | 21
kilogram (kg) | -0.19 [-0.40 to 0.02]

21. Secondary Outcome: Change in Knee Strength
Description: Humac isokinetic dynamometer to measure isokinetic power and isometric strength of knee flexors extensors
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: change in maximum kilograms
Arm/Group | Intervention
Number analyzed (Participants) | 21
change in maximum kilograms
  Right knee flexors | 3.34 [-0.74 to 7.41]
  Left knee flexors | -0.84 [-6.36 to 4.69]
  Right knee extensors | 9.99 [1.80 to 18.18]
  Left knee extensors | 9.86 [0.40 to 19.33]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Baseline through the 12 week follow-up visit (an overall total of 12 weeks).
Description: Lab team members who became aware of any adverse event or unanticipated problems related to the study were to notify the PIs immediately. All adverse events and study-related safety events were collected by the study team. Aggregated unanticipated problems and adverse events were reviewed on a monthly basis, or more often if urgent matters arose.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
This was a single arm study so it is not known how HIIT compares to other exercise approaches or interventions for the management of knee OA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03281668/Prot_SAP_000.pdf